CLINICAL TRIAL: NCT07081646
Title: A Phase 1b/2 Study of AZD0120 (Also Known as GC012F), a Chimeric Antigen Receptor T Cell Therapy Targeting CD19 and B Cell Maturation Antigen in Participants With Relapsed or Refractory AL Amyloidosis.
Brief Title: A Phase 1b/2 Study of CAR T Cell Therapy Targeting CD19 and BCMA in Participants With Relapsed or Refractory AL Amyloidosis.
Acronym: ALACRITY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D831AC00001; AZD0120-AL-201 (Registry Identifier: Alexion)
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Relapsed AL Amyloidosis; Refractory AL Amyloidosis; Light Chain Amyloidosis; Amyloidosis
Keywords: AZD0120; Amyloidosis; AL Amyloidosis; CAR-T; Cell Therapy
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD0120 (Experimental): Participants will receive weight-based dose of AZD0120.
  Interventions: Drug: AZD0120

INTERVENTIONS:
Drug: AZD0120 — Participants will receive AZD0120 via intravenous (IV) infusion.

SUMMARY:
Open-label Phase 1b/2 study with primary objective of this study is to evaluate the safety, tolerability and efficacy of AZD0120 in participants with light chain (AL) amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histopathological diagnosis of AL amyloidosis
* One or more organs currently or historically impacted by AL amyloidosis according to consensus guidelines
* Measurable hematologic disease: dFLC > 20 mg/L or serum M-protein > 5g/L
* Relapsed disease or refractory disease defined as a need for additional therapy after at least 1 line of anti-plasma cell-directed therapy.
* ECOG performance status of 0 to 1
* Must be able and willing to adhere to the study visit schedule and other protocol requirements
* Women of child-bearing potential (WCBP) must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study.

Exclusion Criteria:

* Have any other form of amyloidosis other than AL amyloidosis
* Mayo Stage IIIb AL amyloidosis
* Oxygen saturation < 95% on room air
* Systolic blood pressure <100mmHg
* NYHA class III or IV
* Extensive GI involvement with evidence of active GI bleeding/risk of bleeding as determined by Investigator
* Prior therapies:

  1. CAR T cell therapy directed at any target
  2. Prior BCMA-targeting therapy
  3. Prior treatment with any FDA approved or investigational T cell engaging therapies (including T cell-directed bispecific or trispecific therapies) at any target within the last 6 months.
* Toxicity from previous anti-cancer or anti-PC-directed therapy did not resolve to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy.
* Active plasma cell leukemia at the time of screening
* Symptomatic multiple myeloma (defined as clonal bone marrow plasma cells ≥10% plus at least one myeloma-defining event per IMWG 2014)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-08-15 (Estimated); Study Completion 2030-12-19 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of Participants With incidence and severity of Treatment-emergent Adverse Events | Through study completion, a minimum of 6 months
Phase 2: Proportion of Participants Experiencing a Complete Response | Through study completion, a minimum of 6 months

SECONDARY OUTCOMES:
Phase 1b: Levels of AZD0120 in blood over time in participants with AL amyloidosis | Through study completion, a minimum of 6 months
Phase 2: Percentage of participants achieving hematologic response | Through study completion, a minimum of 6 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Research Site, Phoenix, Arizona
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Nashville, Tennessee
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR